CLINICAL TRIAL: NCT06898684
Title: Medulloblastoma Online Video-based Exercise Pilot Study (MOVE)
Brief Title: Medulloblastoma Online Video-based Exercise Pilot Study
Acronym: MOVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aron Onerup (Other Government)
Collaborators: Göteborg University (Other); Uppsala University (Other); Region Västerbotten (Other Government); Region Stockholm (Other Government); Region Östergötland (Other); Region Skane (Other); Technical University of Munich (Other); Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor-Investigator, Aron Onerup, Principal investigator, Vastra Gotaland Region
Organization: Vastra Gotaland Region (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MOVE pilot
Record Dates: First submitted 2025-03-13; First posted 2025-03-27 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Medulloblastoma, Childhood
Keywords: exercise; rehabilitation; medulloblastoma
MeSH Terms: conditions — Medulloblastoma; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise (Experimental): Video-supervised exercise, offered three times per week for 12 weeks, followed by behavioral support towards incorporating physical activity into daily life for an additional 12 weeks.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Moderate-high intensity exercise, with three sessions per week during 12 weeks. Includes both aerobic and resistance training and will also include exercises that strengthen coordination and balance.

SUMMARY:
In this study, the investigators test whether it is possible to deliver an exercise intervention via video meetings to children and adolescents who have completed therapy for medulloblastoma. The exercise sessions will be individualized and offered three times weekly during 12 weeks.

DETAILED DESCRIPTION:
Tumors of the central nervous system (CNS) represent 25-30% of all cases of pediatric cancer in Sweden. The survival for children with a brain tumor has improved over the last years. The 5-year overall survival rate is now 70%, resulting in a growing number or survivors every year. Malignant brain tumors typically have a poor prognosis, and curative treatment usually requires a combination of neurosurgery, chemotherapy and/or radiotherapy. For the survivors, the cure often comes at the cost of long-term side effects. Finding effective ways to mitigate the long-term side effects after childhood brain tumor is important, since they can severely impact the survivors´ daily life.

There is growing evidence that physical exercise is beneficial to cognition and improves cardiorespiratory fitness and motor function. It appears to be important that interventions start early, within 1-2 years after radiotherapy. For this to be feasible in international multicenter trials, the intervention and outcome assessments will need to be delivered remotely. Whether this is feasible in children treated for medulloblastoma is not known.

The investigators will perform a pilot study to provide pivotal information on whether exercise training can be remotely delivered in the home environment in children treated for medulloblastoma. This will take exercise training from an interesting research concept into a scalable intervention that can be offered regardless of geographic location of the patient. The study will further define the validity and feasibility of in-home outcome assessments of cardiorespiratory, muscular fitness and motor function in children treated for medulloblastoma. If shown feasible, this will work as a proof-of-concept and lead the way for including physical activity intervention in other childhood cancer treatment protocols as well. The results from this study will also enable the researchers to proceed in the planning of the first exercise intervention to be included upfront in an international childhood cancer treatment protocol, the upcoming Pan-European treatment protocol for standard-risk medulloblastoma in children (SIOP-MB6).

ELIGIBILITY:
Inclusion Criteria: Completed therapy for medulloblastoma, including craniospinal radiation therapy, within 36 months before study entry.

-

Exclusion Criteria: Inability to walk without support. Progressive disease.

-

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-12-09 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the remote assessment and a digitally delivered exercise intervention | From enrollment to the end of exercise at 12 weeks and then for prolonged support for another 12 weeks.
  The researchers will test the feasibility of delivering the exercise intervention via video, defined as:
  1. Adherence to the intervention by number of completed intervention sessions Acceptable level: ≥70% adherence at 6 months.
  2. Data collection - feasibility of outcome measures Criteria: ≥ 90% of video-based measurements can be conducted according to protocol. ≥ 80% of PROM assessments can be completed as planned.
  3. Safety Documentation of adverse events (all occurring and documented adverse events associated with the intervention will be recorded in accordance with the Common Terminology Criteria for Adverse Events (CTCAE), version 5.0.).
  4. Acceptance and perceived usefulness Criterion: Qualitative analysis of interviews shows that the intervention is perceived as meaningful, feasible, and not too burdensome.
  5. Technical aspects Criterion: ≥ 90% of participants can complete video sessions without major technical problems, beginning after the first three sessions.

SECONDARY OUTCOMES:
Handgrip strength | Change from baseline, until 3 and 12 months.
  Measured with a hand dynamometer
Physical activity | Change from baseline, until 1.5, 3, 6, and 12 months.
  Activity counts per day, registered with accelerometry (Fibion Sens)
Patient-reported quality of life | Change from baseline, until 3 and 12 months.
  Measured with Patient-Reported Outcomes Measurement Information System (PROMIS)-25.
Motor function | Change from baseline, until 3 and 12 months.
  Assessed with the brief ataxia rating scale (BARS), higher numbers indicate worse outcomes.
Cardiorespiratory fitness | Change from baseline, until 3 and 12 months.
  Assessed with the 3-min step in place test
Epigenetic age acceleration | Change from baseline, until 3 and 12 months.
  Epigenetic age will be determined from DNA methylation analyses of DNA extracted from saliva samples.
Feasibility of the outcome measures | 12 weeks
  The researchers will develop the outcome assessments battery by removing outcome assessments that are not feasible through video.
Cognitive function | Change from baseline to 12 weeks and 12 months.
  Patient-Reported Outcomes Measurement Information System (PROMIS) cognitive function 7a.
Lower limb strength | Change from baseline until 3 and 12 months.
  We will assess lower limb strength with the five repetition sit-to-stand test, assessed with the number of seconds to perform the test. The same chair will be used across all time points.

CONTACTS AND LOCATIONS:
Locations (2):
- Technical University Munich, München, Germany
- Queen Silvia C hildren´s Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No
This is a small feasibility study and will not generate data that will be meaningful to share.